CLINICAL TRIAL: NCT00001234
Title: Retroviral-Mediated Transfer and Expression of Glucocerebrosidase and Ceramidtrihexosidase (a-Galactosidase A) cDNA's in Human Hematopoietic Progenitor Cells
Brief Title: Gene Therapy for Gaucher's and Fabry Disease Using Viruses and Blood-Forming Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 880019; 88-N-0019
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-04

CONDITIONS: Gaucher's Disease
Keywords: Bone Marrow; Retroviral-Mediated Gene Transfer; Hematopoietic Progenitor Cell
MeSH Terms: conditions — Gaucher Disease

INTERVENTIONS:
Genetic: human glucocerebrosidase cDNA

SUMMARY:
Gaucher's disease is a lysosomal storage disease resulting from glycocerebroside GLUCOCEREBROSIDE (1) accumulation in macrophages due to a genetic deficiency of the enzyme glucocerebrosidase. It may occur in patients of all ages. The most severe form, Type 2 Gaucher's Disease occurs in infants who die in the first years of life (with rapidly progressive neurologic deterioration). The condition is passed from generation to generation through autosomal recessive inheritance.

Fabry's disease isa genetic disorder (X-linked recessive) due to the absence of the enzyme a-galactosidase A. The disease is characterized by abnormal collections of glycolipids in cells (histiocytes) within blood vessel walls, tumors on the thighs, buttocks, and genitalia(2) decreased sweating, tingling sensations in the extremities, and cataracts. Patients with Fabry's disease die from complications of the kidney, heart, or brain.

Both conditions are caused by the absence of specific enzymes (3). Patients with these conditions are missing (3) or have defective genes needed for the normal production of these enzymes. Studies on the blood-forming cells in bone marrow have lead to gene therapies using retroviruses as vehicles to carry and insert working genes into abnormal or diseased cells.

This study is designed to measure the safety and effectiveness of transferring working copies of genes responsible for making missing enzymes into the cells of patients with Gaucher's or Fabry disease.

DETAILED DESCRIPTION:
This protocol was developed in order to obtain bone marrow stem cells for ex vivo transduction with retroviruses containing the human glucocerebrosidase gene. We continue to enter a small number of patients to this protocol each year. Studies with the bone marrow hematopoietic progenitor cells have enabled us to identify the most effective retroviral construct currently available in order to carry out gene therapy trials in patients with Gaucher's disease. The data revealed that a comparatively simple retroviral construct containing human glucocerebrosidase cDNA driven by the MoLV promoter is highly effective. We have obtained approval and initiated a Phase I safety and gene marking investigation in patients with Type I Gaucher's Disease.

ELIGIBILITY:
Normal and patient volunteers.

Individuals with platelet counts less than 40,000/ul, PT greater than 15 seconds, or PTT greater than 40 seconds will not undergo bone marrow aspiration.

Individuals with hematologic disorders other than Gaucher Disease, Fabry Disease, or mild iron deficiency will not undergo bone marrow aspiration.

HIV positive individuals will be excluded from participating.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 1988-01; Study Completion 2002-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fink JK, Correll PH, Perry LK, Brady RO, Karlsson S. Correction of glucocerebrosidase deficiency after retroviral-mediated gene transfer into hematopoietic progenitor cells from patients with Gaucher disease. Proc Natl Acad Sci U S A. 1990 Mar;87(6):2334-8. doi: 10.1073/pnas.87.6.2334. PMID 2315324
- [Background] Medin JA, Migita M, Pawliuk R, Jacobson S, Amiri M, Kluepfel-Stahl S, Brady RO, Humphries RK, Karlsson S. A bicistronic therapeutic retroviral vector enables sorting of transduced CD34+ cells and corrects the enzyme deficiency in cells from Gaucher patients. Blood. 1996 Mar 1;87(5):1754-62. PMID 8634421
- [Background] Dunbar C, Kohn D. Retroviral mediated transfer of the cDNA for human glucocerebrosidase into hematopoietic stem cells of patients with Gaucher disease. A phase I study. Hum Gene Ther. 1996 Jan 20;7(2):231-53. doi: 10.1089/hum.1996.7.2-231. PMID 8788174